CLINICAL TRIAL: NCT03932058
Title: Establishment of New Molecular Prototyping Based on Proteomics for Predicting Osteosarcoma Chemotherapy Response and Risk of Recurrence
Brief Title: Proteomics Research of Osteosarcoma
Acronym: PROS001
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Principal Investigator, Zhaoming Ye, Professor, Second Affiliated Hospital, School of Medicine, Zhejiang University
Other Study IDs: PR-OS-001
Record Dates: First submitted 2019-04-26; First posted 2019-04-30 (Actual); Last update posted 2019-05-02 (Actual); Status verified 2019-04

CONDITIONS: Osteosarcoma; Proteomics
MeSH Terms: conditions — Osteosarcoma | interventions — Drug Therapy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- osteosarcoma
  Interventions: Drug: Chemotherapy
- chondrosarcoma
- enchondroma

INTERVENTIONS:
Drug: Chemotherapy — all osteosarcoma patients will give regular chemotherapy for osteosarcoma, the protocol is the same as Methotrexate+Doxorubicin+Cisplatin.
  Groups: osteosarcoma

SUMMARY:
Retrospectively collected 400 cases of clinical data and pathological paraffin specimens of osteosarcoma, chondrosarcoma (control) and endogenous chondroma (control) in our hospital from 2008 to 2014, combined with high-pressure cycle-satellite scanning mass spectrometry (PCT-SWATH) Molecular typing of osteosarcoma and prediction of targeted therapy, the establishment of a new molecular classification based on proteomics for osteosarcoma to predict the chemotherapy response and recurrence risk of osteosarcoma. Clinical osteosarcoma patients include as many types as possible: pre-chemotherapy, post-chemotherapy, recurrence, and metastasis. The study did not involve vulnerable groups, and it was taken as a postoperative wax specimen for patients, which had no health, life and other effects on patients. Study application exemption from informed consent.

ELIGIBILITY:
Inclusion Criteria:

* all osteosarcoma patients in our hospital
* received Methotrexate+Doxorubicin+Cisplatin protocol chemotherapy

Exclusion Criteria:

* non-chemotherapy patients
* bio-specimen not completed

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-09-01 (Estimated); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
proteomics changes | 2 years
  Study of changes in proteomes in tumor cells by high-throughput proteomics analysis

CONTACTS AND LOCATIONS:
Overall Officials: zhaoming Ye, Prof., Principal Investigator — 2nd Affiliated Hospital Of Zhejiang University
Locations (1):
- 2nd Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No